CLINICAL TRIAL: NCT06063499
Title: Healthy Minds Program for Veterans With Opioid Use Disorder on Buprenorphine Maintenance Treatment: A Pilot Study
Brief Title: HMP for Addictions Study
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: prioritizing other opportunities
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Center for Healthy Minds (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2024-0247; SMPH/PSYCHIATRY/PSYCHIATRY (Other: UW Madison); Protocol Version 6/30/23 (Other: UW Madison)
Record Dates: First submitted 2023-09-20; First posted 2023-10-02 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Opioid Use Disorder; Opioid Use; Buprenorphine Dependence
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 6 weeks of sessions (Experimental): Participants will be asked to attend 6 2-hour weekly in-person sessions
  Interventions: Behavioral: Healthy Minds Program for Addictions

INTERVENTIONS:
Behavioral: Healthy Minds Program for Addictions — The Healthy Minds Program for Addictions is a 6-week, hybrid version of the original Healthy Minds Program (HMP), in which all lessons are adapted from the original lessons available in the app and delivered exclusively in person over weekly group sessions. The HMP has >100 guided audio practices that address 4 constituents of wellbeing: awareness, connection, insight, and purpose. Study participants will have access to specific practices from the HMP that are particularly relevant to the needs of populations with substance use disorders and trauma.

SUMMARY:
The goal of this clinical trial is to see whether the Healthy Minds Program for Addictions could be used to help veterans with moderate-severe opioid use disorder and post-traumatic stress disorder stay on buprenorphine maintenance treatment.

Participants will be asked to complete a six-week program consisting of 6 weekly, 2-hour in-person group sessions, as well as assessments before the start of the sessions.

DETAILED DESCRIPTION:
This is a 6-week, single-arm, single-center pilot study of the acceptability and efficacy of an adaptation of the Healthy Minds Program for Veterans with opioid use disorder on buprenorphine maintenance treatment.

Following the Screening Visit, eligible subjects will complete 6 in-person sessions over the course of 2 months. The first session will be an introductory session introducing the basics of the program. After the introductory session, there will be four weekly sessions, each dedicated to a different domain of the program - awareness, connection, insight, and purpose. Participants will be encouraged to practice daily anywhere from 5 to 30 minutes from a set of practices that will be available to them on a password protected website. The intervention will end with a closing session where participants will have the opportunity to reflect on their experience of the program and share feedback. Weekly sessions will be held in person and will be facilitated by an MD, PhD Psychiatrist and Neuroscientist with 8 years of mindfulness practice together with a certified Peer Support Specialist.

ELIGIBILITY:
Inclusion Criteria:

* Individuals at least 18 years of age
* English-speaking
* Veterans
* Ability to understand and willingness to sign a written informed consent document
* Have access to a smartphone, tablet, or computer with internet connection to access recordings for home practice
* Ability and willingness to attend all 6 session of the study, and to complete all assessment questionnaires
* Verified Post-Traumatic Stress Disorder (PTSD) according to DSM-5 criteria
* On buprenorphine maintenance treatment for Opioid use disorder (OUD) for a minimum of 3 months

Exclusion Criteria:

* Regular daily meditation practice for past 6 months or regular weekly meditation practice for past 12 months
* Attended a meditation retreat or a yoga/body practice retreat with a significant meditation component
* Previous use of Healthy Minds Program app
* Current suicidal intent and/or high self-injury risk, as determined from the interview
* Current psychopathology that interferes with study participation as assessed by interview

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-05 (Estimated); Primary Completion 2025-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Retention in treatment | Through study completion, up to 4 months
  Number of participants who complete all 6 sessions, as measured through actual attendance.
Change in predictors of relapse and recovery | Baseline, 3 weeks, 6 weeks
  The Brief Addiction Monitor (BAM) is a 17-item, multidimensional, progress-monitoring instrument for patients in treatment for a substance use disorder (SUD). The BAM includes items that assess risk factors for substance use (scores 0-24, higher scores meaning more risk), protective factors that support sobriety (scores 0-24, higher scores meaning more protection), and drug and alcohol use (scores 0-12, higher scores meaning more use). The BAM produces composite scores for the three aforementioned domains.

SECONDARY OUTCOMES:
Change in psychological distress - perceived stress | Baseline, 3 weeks, 6 weeks
  Stress will be measured using the 10-item NIH Perceived Stress Scale. Each question is scored from 0 (never) to 5 (very often). The total score ranges from 0 to 40, with higher scores indicating higher levels of stress.
Change in psychological distress - anxiety and depression | Baseline, 3 weeks, 6 weeks
  Anxiety and depression will be measured using the Patient Reported Outcomes Measurement Information Systems (PROMIS) Anxiety and Depression scales. The investigators will use the computer adaptive version of both measures which have a mean of 50 and a standard deviation of 10. A composite will be computed by average across T-scores. T-scores range from 10 to 90 with higher scores indicating higher depression or anxiety.
Change in PTSD symptoms | Baseline, 3 weeks, 6 weeks
  PTSD symptoms will be measured by the PTSD Checklist for Diagnostic and Statistical Manual of Mental Disorders (PCL-5). The PCL-5 uses a 5-point Likert scale ranging from 0-4 for each symptom. Respondents rate how bothered they have been by each item in the past month. The items are summed to provide a total severity score ranging from 0-80. Higher scores indicate a higher level of symptoms.
Change in well-being | Baseline, 3 weeks, 6 weeks
  Well-being will be measured using the 17-item Healthy Minds Index (HMI). The HMI assesses qualities trained in the HMP app (awareness, connection, insight, purpose). It is scored on a 0- to 4-point Likert scale where 0 = a low amount (e.g., never, not at all, none of the time) and 4 = a higher amount (e.g., always, to the highest degree, all of the time) of a particular quality.

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Juergens, MD, Principal Investigator — University of Wisconsin, Madison

IPD SHARING:
Plan to Share IPD: No